CLINICAL TRIAL: NCT05932017
Title: Comparison of Gingival Flap Procedure Using Conventional Surgical Loupes vs. Videoscope for Visualization. A Pilot Study
Brief Title: Comparison of Gingival Flap Procedure Using Conventional Surgical Loupes vs. Videoscope for Visualization
Status: Enrolling by invitation | Type: Observational
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB2022-1044
Record Dates: First submitted 2023-03-27; First posted 2023-07-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Periodontal Diseases; Periodontal Pocket; Periodontitis; Periodontal Inflammation; Periodontal Attachment Loss; Periodontal Bone Loss; Surgery
Keywords: videoscope
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; Periodontitis; Periodontal Attachment Loss; Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gingival crevicular fluid (collected through commercially available paper points) and saliva (collected through a tube) will be analyzed for detection of bacterial species. Analysis of saliva and gingival crevicular fluid is standard regimen and commercially available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients receiving routine, pre-diagnosed, standard of care procedures.: Single cohort of patients receiving previously prescribed treatment. The only variable will be the modality of visualization utilized on each side of the mouth during the surgical procedure.

SUMMARY:
This study is being performed to compare different methods of visualization during routine gum surgery. The gum surgery is standard of care. This study will compare the use of a small camera (videoscope) in conjunction with magnification glasses during surgery vs. surgery only using magnification glasses. Both methods are routinely used and are standard of care methods of visualization. The small camera (videoscope) is a device which allows us to see the area under high magnification and projects live video feed on a computer screen.

The study is a split-mouth design pilot study. The patients are only receiving treatment that was previously diagnosed prior to entering the study. The treatment performed is standard treatment that fits in the routine standard of care. No interventional treatment is being performed. The only difference is the method of visualization/observation by the practitioner used during the surgical procedure. One side of the mouth will be treated with just loupes while the other side of the mouth will be treated with loupes and the videoscope.

DETAILED DESCRIPTION:
It is well known that tartar makes at-home oral hygiene care more difficult. The plaque and bacteria that accumulate on tartar are considered the primary factors contributing to gum disease. Conventional gum surgery is commonly performed using loupes (magnification glasses). The use of a videoscope, a handheld miniature camera, allows for greater visualization during surgery. While the debris on the root surface of teeth is not visible with loupes, it is easily observed when the root surface is visualized with the high magnification of the videoscope. The videoscope allows for up to 40x magnification to visualize underneath the gumline. The use of loupes and the videoscope are methods of visualization that are standard of care at the Texas A&M College of Dentistry.

This study is being performed to compare different methods of visualization during routine gum surgery. The gum surgery is standard of care. This study will compare the use of the videoscope in conjunction with loupes during surgery vs. surgery only using loupes. No aspect of this study is investigational, however, bacterial samples will be collected from the patients at multiple time points to assess outcomes. The collection of bacterial samples for research will be conducted through paper points and an oral rinse. These methods are well-established methods of data collection.

Data will be sent to OralDNA labs for analysis. A special contract is required between the school and the company as they will be paid for the services rendered.

Hypothesis: Does the use of the videoscope in conjunction with loupes, as compared to only using loupes for visualization during surgery, have a positive effect (i.e. reduced inflammation and active disease) on the outcomes of gum surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are treatment planned for open flap debridement in two or more quadrants
* age >18 years old
* Stage III periodontitis diagnosis
* Probing depths ≥5mm with bleeding on probing

Exclusion Criteria:

* systemic disease affecting bone metabolism
* current smokers
* diabetes
* pregnant women
* adults unable to consent
* prisoners
* previous or current bisphosphonate use
* recent joint replacement requiring prophylactic antibiotics
* teeth that necessitate and undergo osseous recontouring (shaping of the bone) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be identified at the Texas A&M University dental school clinic.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Probing Depth (in millimeters) | baseline
  The distance from the soft tissue (gingiva or alveolar mucosa) margin to the tip of the periodontal probe during usual periodontal diagnostic probing. The health of the attachment apparatus can affect the measurement. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
  The instrument used to measure the probing depth is the periodontal probe. The periodontal is a calibrated probe used to measure the depth and determine the configuration of a periodontal pocket. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
Clinical Attachment Level (in millimeters) | baseline
  The distance from the cemento-enamel junction to the tip of the periodontal probe during usual periodontal diagnostic probing. The health of the attachment apparatus can affect the measurement. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
  The instrument used to measure the clinical attachment level is the periodontal probe. The periodontal is a calibrated probe used to measure the depth and determine the configuration of a periodontal pocket. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
Bleeding on Probing (yes or no) | baseline
  Bleeding is observed or not observed around each of 6 surfaces for each individual tooth following the gentle probing into the gingiva to obtain the probing depth measurements (see definition of periodontal probing). Gingival bleeding indicates the presence of inflammation. Bleeding on probing is a standard of care observation/finding and clinical sign that indicates the presence of inflammation and the progression of periodontal disease.
Probing Depth (in millimeters) | These will be collected at 3 months post-surgery.
  The distance from the soft tissue (gingiva or alveolar mucosa) margin to the tip of the periodontal probe during usual periodontal diagnostic probing. The health of the attachment apparatus can affect the measurement. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
  The instrument used to measure the probing depth is the periodontal probe. The periodontal is a calibrated probe used to measure the depth and determine the configuration of a periodontal pocket. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
Clinical Attachment Level (in millimeters) | These will be collected at 3 months post-surgery.
  The distance from the cemento-enamel junction to the tip of the periodontal probe during usual periodontal diagnostic probing. The health of the attachment apparatus can affect the measurement. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
  The instrument used to measure the clinical attachment level is the periodontal probe. The periodontal is a calibrated probe used to measure the depth and determine the configuration of a periodontal pocket. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
Bleeding on Probing | These will be collected at 3 months post-surgery.
  Bleeding is observed or not observed around each of 6 surfaces for each individual tooth following the gentle probing into the gingiva to obtain the probing depth measurements (see definition of periodontal probing). Gingival bleeding indicates the presence of inflammation. Bleeding on probing is a standard of care observation/finding and clinical sign that indicates the presence of inflammation and the progression of periodontal disease.
Probing Depth (in millimeters) | These will be collected at 6 months post-surgery.
  The distance from the soft tissue (gingiva or alveolar mucosa) margin to the tip of the periodontal probe during usual periodontal diagnostic probing. The health of the attachment apparatus can affect the measurement. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
  The instrument used to measure the probing depth is the periodontal probe. The periodontal is a calibrated probe used to measure the depth and determine the configuration of a periodontal pocket. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
Clinical Attachment Level (in millimeters) | These will be collected at 6 months post-surgery.
  The distance from the cemento-enamel junction to the tip of the periodontal probe during usual periodontal diagnostic probing. The health of the attachment apparatus can affect the measurement. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
  The instrument used to measure the clinical attachment level is the periodontal probe. The periodontal is a calibrated probe used to measure the depth and determine the configuration of a periodontal pocket. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
Bleeding on Probing | These will be collected at 6 months post-surgery.
  Bleeding is observed or not observed around each of 6 surfaces for each individual tooth following the gentle probing into the gingiva to obtain the probing depth measurements (see definition of periodontal probing). Gingival bleeding indicates the presence of inflammation. Bleeding on probing is a standard of care observation/finding and clinical sign that indicates the presence of inflammation and the progression of periodontal disease.
Probing Depths (in millimeters) | These will be collected at 1 year post-surgery.
  The distance from the soft tissue (gingiva or alveolar mucosa) margin to the tip of the periodontal probe during usual periodontal diagnostic probing. The health of the attachment apparatus can affect the measurement. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
  The instrument used to measure the probing depth is the periodontal probe. The periodontal is a calibrated probe used to measure the depth and determine the configuration of a periodontal pocket. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
Clinical Attachment Level (in millimeters) | These will be collected at 1 year post-surgery.
  The distance from the cemento-enamel junction to the tip of the periodontal probe during usual periodontal diagnostic probing. The health of the attachment apparatus can affect the measurement. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
  The instrument used to measure the clinical attachment level is the periodontal probe. The periodontal is a calibrated probe used to measure the depth and determine the configuration of a periodontal pocket. (Definition from the American Academy of Periodontology Glossary of Periodontal Terms).
Bleeding on Probing | These will be collected at 1 year post-surgery.
  Bleeding is observed or not observed around each of 6 surfaces for each individual tooth following the gentle probing into the gingiva to obtain the probing depth measurements (see definition of periodontal probing). Gingival bleeding indicates the presence of inflammation. Bleeding on probing is a standard of care observation/finding and clinical sign that indicates the presence of inflammation and the progression of periodontal disease.

SECONDARY OUTCOMES:
Bacterial Species Identification | These will be collected at the initial visit
  Fluid from just underneath the subject's gums will be collected using a using a commercially available test (paper strip). The strip will be analyzed for bacteria. Minimal discomfort is associated with this procedure. The bacterial sampling is not routinely done in our clinic and considered to be a research only procedure. The test samples will be analyzed by OralDNA® Labs.
Bacterial Species Identification | These will be collected at 3 months post-surgery.
  Fluid from just underneath the subject's gums will be collected using a using a commercially available test (paper strip). The strip will be analyzed for bacteria. Minimal discomfort is associated with this procedure. The bacterial sampling is not routinely done in our clinic and considered to be a research only procedure. The test samples will be analyzed by OralDNA® Labs.
Bacterial Species Identification | These will be collected at 6 months post-surgery.
  Fluid from just underneath the subject's gums will be collected using a using a commercially available test (paper strip). The strip will be analyzed for bacteria. Minimal discomfort is associated with this procedure. The bacterial sampling is not routinely done in our clinic and considered to be a research only procedure. The test samples will be analyzed by OralDNA® Labs.
Bacterial Species Identification | These will be collected at 1 year post-surgery.
  Fluid from just underneath the subject's gums will be collected using a using a commercially available test (paper strip). The strip will be analyzed for bacteria. Minimal discomfort is associated with this procedure. The bacterial sampling is not routinely done in our clinic and considered to be a research only procedure. The test samples will be analyzed by OralDNA® Labs.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Parra Carrasquer, DDS, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University School of Dentistry, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT05932017/ICF_000.pdf